CLINICAL TRIAL: NCT01287455
Title: The Effect of Vitamin D Replacement on Airway Reactivity, Allergy and Inflammatory Mediators in Exhaled Breath Condensate in Vitamin D Deficient Asthmatic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 483 CTIL; Vitamin D
Record Dates: First submitted 2011-01-30; First posted 2011-02-01 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Asthma; Vitamin D Deficiency
Keywords: Asthma; Vitamin D; airway reactivity; metacholine challenge test
MeSH Terms: conditions — Asthma; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- vitamin D (Active Comparator): vitamin D deficient asthmatic patients receiving vitamin D supplement
  Interventions: Drug: Vitamin D3 as "BABY D3"
- placebo (Placebo Comparator): vitamin D deficient asthmatic patients receiving placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Vitamin D3 as "BABY D3" — drops, 70 drops (= 14000 units), once weekly for 6 weeks
  Arms: vitamin D
Other: placebo — drops, 70 placebo drops, once weekly for 6 weeks
  Arms: placebo

SUMMARY:
Research Title: The effect of vitamin D replacement on airway reactivity, allergy and inflammatory mediators in exhaled breath condensate in vitamin D deficient asthmatic children.

Introduction: Vitamin D seems to play a role in allergic and asthmatic reactions as an immunomodulator. Asthma disease involves inflammatory process in the lower respiratory tract and airway hyperreactivity.

Aim: To assess the effect of Vitamin D replacement on airway reactivity, and allergy and inflammatory mediators in exhaled breath condensate in vitamin D deficient asthmatic children.

Design: Double blind placebo control prospective study comparing the effect of Vitamin D replacement and placebo on airway reactivity, allergy and inflammatory mediators in exhaled breath condensate in asthmatic pediatric population with vitamin D deficiency.

Participant selection: The study group will consist of pediatric patients (age 6-18 years) followed and treated at the Pediatric Pulmonary Unit at the investigators hospital.

Patients with mild-moderate asthma with low or insufficient vitamin D levels that are currently not receiving anti-inflammatory treatment will be recruited.

Sample size: 60 participants in the two groups (30 receiving Vitamin D and 30 receiving placebo).

Intervention: Vitamin D (14000 units) or placebo will be provided in a similar appearance preparation once weekly for 6 weeks between visit two and three.

Three visits will be conducted. Each subject will undergo evaluation including a respiratory questionnaire (visit 1), methacholine challenge test with determination of PC20 (visit 1 or 2 and visit 3), exhaled nitric oxide (eNO) (visit 2, 3), and exhaled breath condensate (EBC) (visit 2,3). Venous blood will be analyzed for complete blood count + eosinophils (visit 1, 3), IGE levels (visit 1, 3), and Vitamin D levels (visit 1, 3). Prick skin test for inhaled allergens will be performed (visit 2, 3).

Primary end point: Airway reactivity as assessed by methacholine challenge test.

Secondary outcome parameters: All other parameters are the secondary end points.

ELIGIBILITY:
Inclusion Criteria:

* 6-18 years
* Mild-moderate asthma
* No anti inflammatory treatment over the past 2 weeks

Exclusion Criteria:

* Any Chronic Lung Disease
* Febrile Illness in last 2 weeks
* FEV1 < 65% in study day
* Bronchodilators over the past 24 hours prior to each study
* Participation in any other clinical studies over the past 4 weeks

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Metacholine Challenge Test | study visit 1,3 (6wks- 3 months)
  As assessed by methacholine challenge test with determination of PC20.

SECONDARY OUTCOMES:
IGE | study visit 1,3 (6wks- 3 months)
  in peripheral Blood count
CBC | study visit 1,3 (6wks- 3 months)
  in peripheral Blood count
Fractional Exhaled NO | visit study 2,3 (6wks)
  determination of exhaled NO in Exhaled breath
skin tests for inhaled allergens | visit study 2,3 (6wks)
Exhaled breath condensate | visit study 2,3 (6wks)
  R-tubes test

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, Prof., Principal Investigator — Rambam Health Care Campus
Locations (1):
- RAMBAM Health Care Campus, Haifa, Israel, Israel

REFERENCES:
- [Derived] Dabbah H, Bar Yoseph R, Livnat G, Hakim F, Bentur L. Bronchial Reactivity, Inflammatory and Allergic Parameters, and Vitamin D Levels in Children With Asthma. Respir Care. 2015 Aug;60(8):1157-63. doi: 10.4187/respcare.03763. Epub 2015 Apr 21. PMID 25899478